CLINICAL TRIAL: NCT04384445
Title: A Phase I/II Randomized, Double Blinded, Placebo Trial to Evaluate the Safety and Potential Efficacy of Intravenous Infusion of Zofin for the Treatment of Moderate to SARS Related to COVID-19 Infection vs Placebo
Brief Title: Zofin (Organicell Flow) for Patients With COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ZEO ScientifiX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19881
Record Dates: First submitted 2020-05-09; First posted 2020-05-12 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Corona Virus Infection; COVID-19; SARS; Acute Respiratory Distress Syndrome
Keywords: Human Amniotic Fluid; Exosomes; Human
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: The trial has two groups, each with 10 subjects (n=20). All eligible study subjects will be randomized, double blinded, to either the treatment group or placebo group.
Who Masked: Participant, Investigator
Masking Description: Double blind: neither subjects nor the investigators who are assessing the patient are award of the treatment assignment until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zofin Plus Standard Care (Experimental): Participants in this group will receive standard of care plus Zofin on day 0, day 4 and day 8.
  Interventions: Biological: Zofin
- Placebo Plus Standard Care (Placebo Comparator): Participants in this group will receive standard of care plus placebo (Saline) on day 0, day 4 and day 8.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Zofin — Biological: Zofin will be administered intravenously with 1ml, containing 2-5 x 10^11 particles/mL in addition to the Standard Care. The Zofin dose will be diluted in 100 mL of sterile saline at subject's bedside.
  Arms: Zofin Plus Standard Care
Other: Placebo — Other: Placebo Placebo (saline) will be administered intravenously with 1ml in addition to the Standard Care. The Placebo dose will be diluted in 100 mL of sterile saline at subject's bedside.
  Arms: Placebo Plus Standard Care

SUMMARY:
The purpose of this research study is to evaluate the safety and potential efficacy of Intravenous Infusion of Zofin for treatment of moderate to severe Acute Respiratory Syndrome (SARS) related to COVID-19 infection vs Placebo.

DETAILED DESCRIPTION:
A human coronavirus (HCoV-19) has caused the novel coronavirus disease (COVID-19) outbreak worldwide. Common symptoms of COVID-19 include fever, cough, and shortness of breath. The majority of cases result in mild symptoms, but some can progress into pneumonia and multi-organ failure. According to the severity it is divided into mild, normal, severe and critically ill, which is associated with ICU admission and mortality. At present, the standard treatment of COVD-19 patients is oxygen therapy, mechanical ventilation, and medications to maintain blood pressure. As of today, no specific antiviral therapy is available for patients with COVID-19. Immune activation in some patients, and the appearance of cytokine storm syndrome (CSS) is one of the important causes of severe damage to lungs and other organs, which may lead to death. There is an urgent need to develop new interventions to suppress the excessive immune response in a timely manner during the course of disease, protect alveolar function, and reduce lung and systemic organ damage.

Zofin is an acellular, minimally manipulated product, derived from human amniotic fluid (HAF). This product contains over 300 growth factors, cytokines, and chemokines as well as other extracellular vesicles/nanoparticles derived from amniotic stem and epithelial cells. The product contains a mean concentration of 5.24x10^11 particles/mL with a mean mode size of 125.2nm. Surface marker analysis confirmed the presence of exosome associated proteins CD63, CD81, and CD9 in addition to high expression of CD133. The completed sequencing revealed 102 commonly expressed miRNA (with a 100-copy expression minimum). Bioinformatics analysis linked 63 miRNAs to 1216 RNA targets. Major players in the proinflammatory cytokine cascade found to be targeted by miRNA were discovered in Organicell's product include TNF, IL-6, and IL-8. Additionally, a broader array of pro-inflammatory cytokines is also targeted by the collection of miRNA such as FGF2, IFNB1, IGF1, IL36a, IL37, TGF-B2, VEGFA, CCL8, and CXCL12. It has been suggested in published research that inhibition or suppression of this pro-inflammatory cytokine cascade may reduce the severity of symptoms associated with elevated immune response. Furthermore, the miRNA was found to target 148 genes associated with immune response.

The property of Zofin demonstrates the therapeutic potential as a suppressor of cytokine activation for the reduction of COVID-19 infection severity. This study aims to investigate safety and potential efficacy of HAF derived acellular product in subjects suffering form COVID-19 infection with severe acute respiratory syndrome (SARS).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Subjects age > 18 years at the time of signing the Informed Consent Form.
3. Male or Female
4. Must have a clinical diagnosis of COVID-19, with at least one of clinical symptoms (e.g., fever ≥38°C, fatigue, cough) and a positive result by the reverse- transcription polymerase chain reaction (RT-PCR) testing or equivalent.
5. Individuals with moderately to severe COVID-19 symptoms.

   Moderate ARDS according to Berlin Criteria:

   Symptoms include: abnormal chest imaging or any degree of hypoxia requiring supplemental oxygen. Bilateral opacities-not fully explained by effusions, lobar/lung collapse, or nodules. Oxygenation: 100 mm Hg < PaO2/FIO2 </= 200 mm Hg with PEEP >/=5 cm H2O

   Severe ARDS according to Berlin Criteria:

   Symptoms include: abnormal chest imaging or any degree of hypoxia requiring supplemental oxygen. Bilateral opacities-not fully explained by effusions, lobar/lung collapse, or nodules. Oxygenation: PaO2/FIO2 </= 100 mm Hg with PEEP >/= 5 cm H2O
6. Hospitalized and symptomatic (cough, fevers, SOB, or sputum production)
7. Adequate venous access
8. Ability to provide informed consent or an authorized representative can sign the informed consent
9. For female patients only, willingness to use FDA- recommended birth control (http://www.fda.gov/downloads/ForConsumers/ByAu dience/ForWomen/FreePublications/UCM356451.pdf ) until 6 months post treatment.
10. Must agree to comply with all study requirements and be willing to complete all study visits
11. Willingness of study participant to accept this treatment arm, and signed informed consent; Need in- patient admission.

Exclusion Criteria:

1. Intubated or on a ventilator.
2. Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods. Female subjects must undergo a blood or urine pregnancy test at screening and within 36 hours prior to infusion.
3. Inability to perform any of the assessments required for endpoint analysis.
4. Active listing (or expected future listing) for transplant of any organ.
5. Be a solid organ transplant recipient. This does not include prior cell-based therapy (>12 months prior to enrollment), bone, skin, ligament, tendon or corneal grafting. Have a history of organ or cell transplant rejection.
6. History of drug abuse (illegal "street" drugs except marijuana, or prescription medications not being used appropriately for a pre-existing medical condition) or alcohol abuse (≥ 5 drinks/day for ˃ 3 months), or documented medical, occupational, or legal problems arising from the use of alcohol or drugs within the past 24 months
7. Be serum positive for HIV, hepatitis BsAg or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of any infusion associated adverse events | 60 Days
  Safety will be defined by the incidence of any infusion associated adverse events as assessed by treating physician
Incidence of Severe Adverse Events | 60 Days
  Safety will be defined by the incidence of severe adverse events as assessed by treating physician

SECONDARY OUTCOMES:
All Cause Mortality | 60 Days
  Measured at day 60 or at hospital discharge, whichever comes first.
Survival Rate | 60 Days
  Number of participants that are alive at 60 days post first infusion follow up
Cytokine Levels | Day 0, Day 4, Day 8, Day14, Day 21, Day 28
  Measure IL-6, TNF-alpha from serum of blood samples
D-dimer Levels | Day 0, Day 4, Day 8, Day14, Day 21, Day 28
  D-dimer from serum of blood samples methodology using blood samples or nose / throat swab
C-reactive protein Levels | Day 0, Day 4, Day 8, Day14, Day 21, Day 28
  CRP from serum of blood samples
Quantification of the COVID-19 | Day 0, Day 4, Day 8
  Viral load by real time RT methodology using blood samples or nose / throat swab
Improved Organ Failure | Day 30
  Improved organ failure within 30 days, including cardiovascular system, coagulation system, liver, kidney and other extra-pulmonary organs using Sequential Organ Failure Assessment (SOFA) score.
Chest Imaging Changes | Day o, Day 30
  Chest imaging changes for 30 days compare to placebo: 1) Ground-glass opacity,
  - 2) Local patchy shadowing, 3) Bilateral patchy shadowing, and 4) Interstitial abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: George C Shapiro, MD, FACC, Principal Investigator — Chief Medical Officer at Organicell Regenerative Medicine, Inc; Maria Ines Mitrani, MD, PhD, Principal Investigator — Chief Science Officer at Organicell Regenerative Medicine, Inc
Locations (1):
- George C. Shapiro, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No